CLINICAL TRIAL: NCT00595127
Title: A Pilot Trial of Hematopoietic Stem Cell Transplantation for the Treatment of Patients With Fanconi Anemia Lacking a Genotypically Identical Donor, Using Total Body Irradiation, Cyclophosphamide and Fludarabine
Brief Title: Hematopoietic Stem Cell Transplantation for Treatment of Patients With Fanconi Anemia Lacking a Genotypically Identical Donor, Using Total Body Irradiation, Cyclophosphamide and Fludarabine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Miltenyi Biotec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-062
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-06

CONDITIONS: Fanconi Anemia
Keywords: Fanconi; Anemia; Stem Cell; Transplant
MeSH Terms: conditions — Fanconi Anemia; Anemia | interventions — Cyclophosphamide; fludarabine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): This is an open-label single arm study of 131I-8H9, injected intravenously at 10 mCi/1.73 m^2 dose [intended specific activity of ~20 mCi/mg protein] preceded by administration of 50mg/1.73m^2 of unlabeled 8H9.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Radiation: Total body irradiation (TBI)

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide (10mg/kg/day x 4days)
Drug: Fludarabine — Fludarabine (30mg/m^2/day x 5 days)
Radiation: Total body irradiation (TBI) — TBI (450 cGY in a single fraction)

SUMMARY:
The purpose of this research study is to: (1) determine if the combination of low dose total body irradiation, low dose cyclophosphamide and the addition of fludarabine, and a serum to suppress the immune system can allow selected stem cells to take and grow; (2) determine if selected stem cells from the blood or marrow can take and not cause graft-versus-host disease (GvHD), and; (3) evaluate the side effects of the combination of low dose radiation and chemotherapy drugs used for these transplants.

DETAILED DESCRIPTION:
Patients with this disease are born with it and have a fragility of the genes (chromosomes) in all the cells of the body. The fragility of the chromosomes puts patients with FA at high risk for certain cancers. Patients with FA are especially at risk of having diseases of the blood and marrow systems. These include (1) aplastic anemia, a disease where there is a failure of the bone marrow to make blood cells and (2) myelodysplastic syndrome which is represented by a clone of cells of the marrow that becomes "malignant" and stops making adequate numbers of blood cells (it is also called preleukemia.) The progression of the myelodysplastic syndrome will lead to (3) acute leukemia.

If you have Fanconi anemia and suffer from aplastic anemia, myelodysplastic syndrome, or leukemia standard treatment with medications or chemotherapy alone is not likely to cure these problems.

An allogeneic blood or bone marrow (hematopoietic stem cell) transplant can be done to provide you with marrow or blood stem cells from a healthy donor that can develop a normal blood forming system. An allogeneic stem cell transplant can cure the problems of the marrow and blood system. It cannot cure the chromosome fragility of the whole body. When allogeneic stem cell transplants have been done for the treatment of FA using stem cells from donors other than matched siblings, they have been associated with a high risk of rejection of the transplant and of a complication called graft-versus-host disease.

In order for the stem cells to grow and to kill leukemia cells, patients must receive chemotherapy and radiation therapy. This preparation is called cytoreduction. For patients with Fanconi anemia, the standard preparation for stem cell transplantation has been the use of total body irradiation (at a lower dose because of the high risk of side-effects) and a chemotherapy agent called cyclophosphamide (or Cytoxan) also at lower dose. While this has worked well with transplants from matched siblings, it was not enough in transplants from unrelated or cord blood donors and led to a high risk of rejection. In the last few years a medication called fludarabine was used successfully in transplants to give more immunosuppression and kill T-cells. Fludarabine allowed transplants to be done with low risks of rejection, and probably as importantly little risks of added side-effects. The addition of antithymocyte globulin to Total Body Irradiation, cyclophosphamide and fludarabine has made the chances of rejection very low.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis:

* Research participants must be have a diagnosis of Fanconi anemia (confirmed by mitomycin or diepoxybutane [DEB] chromosomal breakage testing).

Hematologic Diagnosis and Status:

* Research participants must have one of the following hematologic diagnoses:

  * Severe Aplastic Anemia (SAA)/Severe Isolated Single lineage Cytopenia
  * Myelodysplastic Syndrome(MDS)
  * Acute leukemia.

HLA-compatible Unrelated volunteer donors:

* Research participants who do not have a related HLA-matched donor but have an unrelated donor who is either matched at all A, B and DRB1 loci or who is mismatched at 1/6 loci (A, B, or DRB1) as tested by DNA analysis, will be eligible for entry on this protocol.

HLA-mismatched Related donors:

* Research participants who do not have a related or unrelated HLA-compatible donor must have a healthy family member who is at least HLA-haplotype identical to the recipient. First degree related donors must have a normal DEB test.
* The donor must be healthy and willing and able (1) to receive a 5 day course of G-CSF and undergo 2 daily leukaphereses, or (2) to undergo general anesthesia and bone marrow donation. In order to undergo a Tcell depletion, a donor should be able to have a volume of 15 ml/Kg of the research participant's body weight harvested safely.

HLA-compatible Cord Blood Units:

* Research participants who do not have a related HLA-matched donor but have an unrelated placental cord blood unit which matched at all A, B and DRB1 loci or who is mismatched at 1/6 or 2/6 loci (A, B, or DRB1) as tested by DNA analysis, will be eligible for entry on this protocol.
* Research participants may be of either gender or any ethnic background.
* Research participants must have a Karnofsky adult, or Lansky pediatric performance scale status > 70%.
* At the time of referral for transplantation, research participants must be in good clinical condition without co-existing medical problems that would significantly increase the risk of the transplant procedure. Research participants must be free of infections at the time of transplant. Research participants must have a life expectancy that is greater than 8 weeks.
* Research participants must have adequate physical function measured by cardiac, Hepatic, Renal, Pulmonary.
* Research participants must be available for follow-up evaluations at 30, 60, 180 days post BMT and yearly for 5 years.

Exclusion Criteria:

* Active CNS leukemic involvement
* Female research participants who are pregnant or breast-feeding
* Active viral, bacterial or fungal infection
* Research participant seropositive for HIV-I/II; HTLV -I/II

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2001-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farid Boulad, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide and Fludarabine: To evaluate a cytoreductive regimen using standard TBI & cyclophosphamide w/ addition of fludarabine, to prepare pts w/ Fanconi anemia for Tcell depleted, allogeneic hematopoietic stem cell transplant
Period: Overall Study
Arm/Group | Cyclophosphamide and Fludarabine
Started | 21
Completed | 11
Not Completed | 10
Not completed — Death | 6
Not completed — Relapsed | 3
Not completed — joined another trial | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide and Fludarabine
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence & Quality of Engraftment & Hematopoietic Reconstitution
Description: Number of patients who engrafted
Time Frame: 8 years
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide and Fludarabine
Number analyzed (Participants) | 21
participants | 19

ADVERSE EVENTS:
Arm/Group | Cyclophosphamide and Fludarabine
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide and Fludarabine (N=21)
Cardiovascular, other (Cardiac disorders) | 1
Diarrhea (PEDS/BMT) (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage, other (Blood and lymphatic system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infection w.out neutropenia (Infections and infestations) | 1
Infection/Feb Neut-Other (Infections and infestations) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide and Fludarabine (N=21)
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Bilirubin (Blood and lymphatic system disorders) | 10
Hemoglobin (Hgb) (Metabolism and nutrition disorders) | 21
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesmia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 14
Hyponatremia (Metabolism and nutrition disorders) | 8
Hypophosphatemia (Metabolism and nutrition disorders) | 11
Leukocytes (Blood and lymphatic system disorders) | 21
Lymphopenia (Blood and lymphatic system disorders) | 21
Neutrophils/gran (Infections and infestations) | 21
Platelets (Blood and lymphatic system disorders) | 21
SGOT (AST) (Metabolism and nutrition disorders) | 9
SGPT (ALT) (Metabolism and nutrition disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes